CLINICAL TRIAL: NCT00322348
Title: An Open-label, Randomised, Parallel Group, Multicentre Study to Compare ZOLADEX 10.8 mg Given Every 12 Weeks With ZOLADEX 3.6 mg Given Every 4 Weeks in Pre-menopausal Women With Oestrogen Receptor Positive Advanced Breast Cancer
Brief Title: Study of Zoladex Given Every 12 Weeks Versus Given Every Month in Advanced Breast Cancer (ABC) Pre-menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D8664C00008; Zoladex ABC Study
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2010-12

CONDITIONS: Advanced Breast Cancer
Keywords: oncology; cancer; breast cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Goserelin

ARMS (2):
- ZOLADEX 10.8 mg (Experimental): ZOLADEX (goserelin acetate) 10.8 mg intramuscular depot for injection every 12 weeks
  Interventions: Drug: Goserelin acetate
- ZOLADEX 3.6 mg (Experimental): ZOLADEX (goserelin acetate) 3.6 mg intramuscular depot for injection every 4 weeks
  Interventions: Drug: Goserelin acetate

INTERVENTIONS:
Drug: Goserelin acetate — 3.6 mg intramuscular depot injection given every 4 weeks
  Other Names: Zoladex®
  Arms: ZOLADEX 3.6 mg
Drug: Goserelin acetate — 10.8 mg intramuscular depot injection given every 12 weeks
  Other Names: Zoladex®
  Arms: ZOLADEX 10.8 mg

SUMMARY:
The primary objective is to evaluate whether Zoladex 10.8 mg (12-weekly) is non-inferior to Zoladex 3.6 mg (4-weekly) in pre-menopausal women with oestrogen receptor positive advanced breast cancer by assessment of progression-free survival at 24 weeks.

Secondary Objectives are to compare the safety and tolerability profile of ZOLADEX 10.8 mg and ZOLADEX 3.6 mg by assessment of adverse events (AEs)and to assess goserelin PK in Japanese and Caucasian participants who have received ZOLADEX 10.8 mg by assessment of goserelin plasma concentration time profiles

Recruitment into the study has been permanently stopped as of 24 December 2007 due to slow recruitment. 98 (vs the planned 260) patients were randomised into the study and will be followed as per protocol for 2 years

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18 years or over with histologically/cytologically-confirmed oestrogen receptor positive (ER +ve) breast cancer
* World Health Organization (WHO) performance status of 0, 1, or 2
* Provided written informed consent

Exclusion Criteria:

* Treatment with tamoxifen or other hormonal therapies as early breast cancer (EBC) adjuvant in the previous 24 weeks
* Received radiotherapy within the past 4 weeks
* History of systemic malignancy other than breast cancer within the previous 3 years
* Estimated survival less than 24 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-04; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Breast Cancer Established Brands Team Medical Science Director, MD, Study Director — AstraZeneca
Locations (14):
- Research Site, Prague, Czechia
- Russia (8):
  - Research Site, Arkhangelsk
  - Research Site, Belgorod
  - Research Site, Kaliningarad
  - Research Site, Kazan, Tatarstan
  - Research Site, Moscow
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Ukraine (5):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Odesa
  - Research Site, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-menopausal women with Oestrogen Receptor Positive Advanced Breast Cancer were recruited between 25th April 2006 and 24th December 2007. 49 participants were randomised to ZOLADEX 10.8 mg and 49 participants were randomised to ZOLADEX 3.6 mg. One participant was randomised to ZOLADEX 3.6 mg but received ZOLADEX 10.8 mg.
Pre-assignment Details: 53 of the151 screened participants were not randomised to treatment groups for the following reasons : 50 participants were incorrectly enrolled (i.e. did not comply with inclusions/exclusion criteria) and a bone scan was not performed for 3 participants.
Period: Overall Study
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Started | 49 | 49
Received Study Treatment | 50 | 48
Completed | 12 (Number of participants completed up to Week 96) | 16 (Number of participants completed up to Week 96)
Not Completed | 37 | 33
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 2
Not completed — Disease Progression | 30 | 25
Not completed — Reasons not specified | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg | Total
Number analyzed (Participants) | 49 | 49 | 98
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (6.45) | 42.6 (6.07) | 42.3 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 27 | 32 | 59
  Black | 0 | 0 | 0
  Oriental | 22 | 17 | 39
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at Week 24
Description: The number of participants for whom neither objective disease progression or death (due to any cause) has been observed at Week 24 over the number of randomised participants x 100.
Time Frame: Objective tumour assessments carried out every 12 weeks (+/- 7 days) until Week 24, and then every 24 weeks (+/- 14 days) until Week 96 or objective progression is confirmed according to Response Evaluation Criteria in Solid Tumours (RECIST).
Measure: Number; unit: Percentage of participants
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 49 | 49
Percentage of participants | 69.4 | 73.5

2. Secondary Outcome: Objective Response Rate (ORR) at Week 24
Description: Number of participants who were objective responders at Week 24 over the number of participants evaluable for response x 100. An objective responder = a participants whose best unconfirmed response is either CR (Complete Response Disappearance of all target lesions) or PR (Partial Response At least a 30% decrease in target lesions)
Time Frame: Response Evaluation Criteria in Solid Tumours (RECIST) tumour assessments carried out every 12 weeks from randomisation until Week 24 in those patients with measurable disease at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 45 | 43
Percentage of participants | 28.9 | 25.6

3. Secondary Outcome: Oestradiol (E2) Serum Concentrations at Week 24
Description: A comparison of mean E2 serum concentrations at timepoint(s) post Day 1 performed using analysis of covariance (ANCOVA), with treatment group, baseline E2 serum concentrations and country as covariates. Data analysed on the log scale; log scale mean and pooled log scale standard deviation from Analysis of Covariance (ANCOVA) presented.
Time Frame: Blood samples for measurement of E2 concentrations collected from all patients at scheduled visits of screening, Day 1 and Weeks 12 and 24 (+/- 7 days). Week 24 data is presented
Measure: Log Mean (Standard Deviation); unit: pmol/L
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 41 | 45
pmol/L | 1.42 (0.99) | 1.49 (0.99)

4. Secondary Outcome: Maximum Plasma Concentration, Cmax (ng/mL)
Description: Maximum plasma concentration, Cmax (ng/mL), derived from analysis of pharmacokinetic (PK) outcomes samples provided only by participants in the PK subgroup set (all of whom received ZOLADEX 10.8 mg)
Time Frame: Blood samples taken at Days 1, 2 and 3, Weeks 4, 12 and 24. Derived from the individual goserelin plasma concentration-time profiles following the first dose of study drug for patients in the pharmacokinetic (PK) subgroup
Population: participants in the pharmacokinetic (PK) subgroup
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 19 | 0
ng/mL | 4.565 [0.501 to 14.000] |

5. Secondary Outcome: Time to Maximum Plasma Concentration, Tmax (Hours)
Description: Time to maximum plasma concentration, Tmax (hours), derived from analysis of pharmacokinetic (PK) outcomes samples provided only by participants in the PK subgroup set (all of whom received ZOLADEX 10.8 mg)
Time Frame: as for outcome 4
Population: participants in the PK subgroup set
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 19 | 0
hours | 1.9 [1 to 24] |

6. Secondary Outcome: Area Under the Plasma Concentration Curve (0-12 Weeks)
Description: Area under the plasma concentration curve (0-12 weeks) derived from analysis of pharmacokinetic (PK) outcomes samples provided only by participants in the PK subgroup set (all of whom received ZOLADEX 10.8 mg)
Time Frame: as for outcome 4
Population: participants in the PK subgroup set
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Number analyzed (Participants) | 19 | 0
ng/mL | 33.021 [9.13 to 73.70] |

ADVERSE EVENTS:
Description: 49 participants were randomised to ZOLADEX 10.8 mg and 49 patients were randomised to ZOLADEX 3.6 mg. One patient was randomised to ZOLADEX 3.6 mg but received ZOLADEX 10.8 mg. therefore 50 participants included in ZOLADEX 10.8 mg and 48 in ZOLADEX 3.6
Arm/Group | ZOLADEX 10.8 mg | ZOLADEX 3.6 mg
Serious Adverse Events (participants affected / at risk) | 2/50 | 3/48
Other Adverse Events (participants affected / at risk) | 39/50 | 37/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZOLADEX 10.8 mg (N=50) | ZOLADEX 3.6 mg (N=48)
Peritonsillar Abscess (Infections and infestations) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Haematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZOLADEX 10.8 mg (N=50) | ZOLADEX 3.6 mg (N=48)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 4
Abdominal Pain (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 0 | 4
Pyrexia (General disorders) | 1 | 4
Asthenia (General disorders) | 1 | 3
Nasopharyngitis (Infections and infestations) | 11 | 5
Respiratory Tract Infection Viral (Infections and infestations) | 3 | 2
Weight Increased (Infections and infestations) | 7 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Headache (Nervous system disorders) | 4 | 3
Amenorrhoea (Reproductive system and breast disorders) | 13 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Hot Flush (Vascular disorders) | 19 | 18

LIMITATIONS AND CAVEATS:
The criteria for non-inferiority were not met for the primary efficacy endpoint (PFS at Week 24). However, since recruitment was terminated prematurely, the study was no longer adequately powered to detect non-inferiority.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents). The only disclosure restriction on the PI is that they cannot disclose or publish any information to do with the trial without consent from AstraZeneca.